CLINICAL TRIAL: NCT01382719
Title: A Placebo-controlled, Randomized, Parallel Group, Dose-finding Trial to Evaluate the Efficacy and Safety of Subcutaneously Administered Bremelanotide in Premenopausal Women With FSAD (Female Sexual Arousal Disorder) and/or HSDD (Hypoactive Sexual Desire Disorder)
Brief Title: Bremelanotide in Premenopausal Women With Female Sexual Arousal Disorder and/or Hypoactive Sexual Desire Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palatin Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PT-141-54
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Female Sexual Arousal Disorder; Hypoactive Sexual Desire Disorder
Keywords: FSAD; HSDD; female sexual dysfunction; FSD; Female Sexual Arousal Disorder; Hypoactive Sexual Desire Disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — bremelanotide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Same formulation as the investigation product but without the active ingredient, provided as pre-filled syringes containing 0.3 mL volume. Subjects will self-administer the placebo by SC injection in the same manner as the investigational product.
  Interventions: Drug: bremelanotide
- bremelanotide arm 1 (Experimental): Low dose: Investigational product: Bremelanotide aqueous solution for subcutaneous (SC) injection, provided as pre-filled syringes containing 0.75 mg in 0.3 mL volume. Subjects will self-administer bremelanotide by SC injection into the anterior thigh or abdomen.
  Interventions: Drug: bremelanotide
- bremelanotide arm 2 (Experimental): Middle dose: Investigational product: Bremelanotide aqueous solution for subcutaneous (SC) injection, provided as pre-filled syringes containing 1.25 mg in 0.3 mL volume. Subjects will self-administer bremelanotide by SC injection into the anterior thigh or abdomen.
  Interventions: Drug: bremelanotide
- bremelanotide arm 3 (Experimental): High dose: Investigational product: Bremelanotide aqueous solution for subcutaneous (SC) injection, provided as pre-filled syringes containing 1.75 mg in 0.3 mL volume. Subjects will self-administer bremelanotide by SC injection into the anterior thigh or abdomen.
  Interventions: Drug: bremelanotide

INTERVENTIONS:
Drug: bremelanotide — Subjects will administer drug on an as needed basis, prior to anticipated sexual activity.
  Investigational product: Bremelanotide aqueous solution for subcutaneous (SC) injection, provided as pre-filled syringes containing 0.75, 1.25, or 1.75 mg in 0.3 mL volume. Subjects will self-administer bremelanotide by SC injection into the anterior thigh or abdomen.
  Placebo: Same formulation as the investigation product but without the active ingredient, provided as pre-filled syringes containing 0.3 mL volume. Subjects will self-administer the placebo by SC injection in the same manner as the investigational product.
  Other Names: PT-141

SUMMARY:
This trial is designed to evaluate the efficacy and safety of 3 fixed dose levels of bremelanotide, administered subcutaneously on an as-needed basis under conditions of home use, for the treatment of female sexual arousal disorder (FSAD), hypoactive sexual desire disorder (HSDD), or mixed FSAD/HSDD in premenopausal women.

ELIGIBILITY:
Inclusion Criteria:

Female, at least 21 years of age, and premenopausal Previously experienced sexual arousal during sexual activity and/or normal level of desire in the past for least 2 years.

Willing to engage in sexual activities Currently in stable relationship with a partner(male or female)for at least 6 months.

If subject has a male sexual partner, has recorded a score of "not impotent" or "minimally impotent" on Single-question Assessment of ED.

For at least 6 months before Screening, has met diagnostic criteria for FSAD, HSDD, or mixed FSAD/HSDD Has a negative serum pregnancy test (hCG) at Screening and, if subject's partner is male, has used a medically acceptable form of contraception for the 3 months before Screening (Visit 1), and is willing to continue for the duration of the trial and 1 month following the last dose of trial drug.

Has a normal pelvic examination. At Screening or documented within 12 months before Screening, has:normal Pap test results with or without history of positive HPV, dysplasia, or ASCUS that has resolved or been treated;Pap test results positive for ASCUS and negative for HPV;Pap test results positive for HPV AND no ASCUS or dysplasia on Pap or condyloma present upon examination.

At Screening and Visit 2, meets all necessary questionnaire scores.

Exclusion Criteria:

Medical condition that is unstable or uncontrolled despite current therapy. History of unresolved sexual trauma or abuse. Pregnant or nursing. Lifelong anorgasmia, vaginismus, sexual pain disorder, sexual aversion disorder, or persistent sexual arousal disorder.

Female sexual dysfunction caused by untreated endocrine disease. Has or has had any of the following: hepatitis C, other infectious hepatitis, infectious blood disorders such as HIV; myocardial infarction;stroke.

Has or has had any of the following within 12 months before Screening:chronic dyspareunia not attributable to vaginal dryness; pelvic inflammatory disease; chronic or complicated UTI, or an active STD other than herpes and condyloma; cervical dysplasia, including LGSIL and HGSIL and/or ASCUS with HPV; significant cervicitis as manifested by mucopurulent discharge from the cervix.

Has had any of the following within 6 months before Screening:≥ 2 outbreaks of genital herpes; occurrence/recurrence of clinically significant condyloma;clinically unstable angina or clinically unstable arrhythmia;significant CNS diseases;AST or ALT concentrations > 3 times the ULN;serum creatinine > 2.5 mg/dL;any other clinically significant abnormal laboratory result.

Has used prohibited medications within the 3 months before Screening:

Has currently active moderate to severe vaginitis or a clinically significant vaginal infection.

Has one or more significant gynecologic conditions . Is taking or has received treatment for psychosis, bipolar disorder, depression, and/or alcohol/substance abuse within 6 months before Screening.

Is currently receiving psychotherapy for the treatment of FSAD and/or HSDD. Has any of the following: Uncontrolled hypertension;Systolic BP of ≥ 140 mm Hg at Screening;Diastolic BP of ≥ 90 mm Hg at Screening; Treatment for hypertension that has changed in the 3 months before Screening.

Had a hysterectomy with bilateral oophorectomy. Had a hysterectomy without bilateral oophorectomy AND meets several other criteria.

Is taking contraceptives that have affected the menstrual cycle or caused amenorrhea AND did not have a normal menstrual cycle before starting the contraceptive medication.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Edelson, MD, FRCPC, Study Director — Palatin Technologies, Inc
Locations (68):
- United States (65):
  - Site 56, Birmingham, Alabama
  - Site 26, Huntsville, Alabama
  - Site 64, Mobile, Alabama
  - Site 45, Chandler, Arizona
  - Site 39, Phoenix, Arizona
  - Site 25, Tucson, Arizona
  - Site 78, Hot Springs, Arkansas
  - Site 16, Jonesboro, Arkansas
  - Site 52, National City, California
  - Site 73, Newport Beach, California
  - Site 80, Sacramento, California
  - Site 12, San Diego, California
  - Site 37, Denver, Colorado
  - Site 40, Lakewood, Colorado
  - Site 8, Avon, Connecticut
  - Site 75, Farmington, Connecticut
  - Site 33, New London, Connecticut
  - Site 32, Washington D.C., District of Columbia
  - Site 10, Aventura, Florida
  - Site 27, Fort Myers, Florida
  - Site 66, Melbourne, Florida
  - Site 61, Orlando, Florida
  - Site 1, West Palm Beach, Florida
  - Site 82, Atlanta, Georgia
  - Site 55, Decatur, Georgia
  - Site 70, Chicago, Illinois
  - Site 54, Peoria, Illinois
  - Site 63, South Bend, Indiana
  - Site 13, Wichita, Kansas
  - Site 48, Lexington, Kentucky
  - Site 57, Zachary, Louisiana
  - Site 9, Baltimore, Maryland
  - Site 60, Rockville, Maryland
  - Site 74, St Louis, Missouri
  - Site 35, Lincoln, Nebraska
  - Site 72, Las Vegas, Nevada
  - Site 24, Las Vegas, Nevada
  - Site 18, New York, New York
  - Site 38, Purchase, New York
  - Site 3, Raleigh, North Carolina
  - Site 47, Winston-Salem, North Carolina
  - Site 23, Beachwood, Ohio
  - Site 69, Canton, Ohio
  - Site 71, Cincinnati, Ohio
  - Site 19, Cleveland, Ohio
  - Site 30, Columbus, Ohio
  - Site 81, Englewood, Ohio
  - Site 2, Eugene, Oregon
  - Site 42, Philadelphia, Pennsylvania
  - Site 77, Pittsburgh, Pennsylvania
  - Site 43, Warwick, Rhode Island
  - Site 58, Greer, South Carolina
  - Site 49, Mt. Pleasant, South Carolina
  - Site 53, Chattanooga, Tennessee
  - Site 59, Corpus Christi, Texas
  - Site 76, Dallas, Texas
  - Site 31, Dallas, Texas
  - Site 17, Houston, Texas
  - Site 62, San Antonio, Texas
  - Site 50, Murray, Utah
  - Site 36, Sandy City, Utah
  - Site 7, Charlottesville, Virginia
  - Site 68, Norfolk, Virginia
  - Site 65, Richmond, Virginia
  - Site 22, Seattle, Washington
- Canada (3):
  - Site 4, North Vancouver, British Columbia
  - Site 41, Barrie, Ontario
  - Site 21, Burlington, Ontario

REFERENCES:
- [Derived] Derogatis LR, Revicki DA, Rosen RC, Jordan R, Lucas J, Spana C. Psychometric validation of the Female Sexual Distress Scale-Desire/Arousal/Orgasm. J Patient Rep Outcomes. 2021 Sep 24;5(1):100. doi: 10.1186/s41687-021-00359-1. PMID 34559353
- [Derived] Clayton AH, Althof SE, Kingsberg S, DeRogatis LR, Kroll R, Goldstein I, Kaminetsky J, Spana C, Lucas J, Jordan R, Portman DJ. Bremelanotide for female sexual dysfunctions in premenopausal women: a randomized, placebo-controlled dose-finding trial. Womens Health (Lond). 2016 Jun;12(3):325-37. doi: 10.2217/whe-2016-0018. Epub 2016 May 16. PMID 27181790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1142 subjects were screened at 69 medical sites in the US and Canada, 612 subjects were enrolled, and 488 subjects entered the single-blind placebo treatment period; 397 were randomized, and 394 were dosed with randomized treatment.
Pre-assignment Details: A total of 91 subjects were not randomized due to failing the resting blood pressure criteria (36), withdrawal of consent (24), being lost to follow-up (9), adverse events (5), non-compliance (5), and other reasons (12).
Groups:
- Placebo: identical formulation without active ingredient
- Bremelanotide Arm 1: low dose 0.75 mg BMT
- Bremelanotide Arm 2: middle dose 1.25 mg BMT
- Bremelanotide Arm 3: high dose 1.75 mg BMT
Period: Overall Study
Arm/Group | Placebo | Bremelanotide Arm 1 | Bremelanotide Arm 2 | Bremelanotide Arm 3
Started | 98 | 100 | 100 | 99
Subjects Not Dosed | 1 | 0 | 1 | 1
Completed | 80 | 81 | 66 | 66
Not Completed | 18 | 19 | 34 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bremelanotide Arm 1 | Bremelanotide Arm 2 | Bremelanotide Arm 3 | Total
Number analyzed (Participants) | 97 | 100 | 99 | 98 | 394
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (7.70) | 37.6 (7.76) | 35.7 (7.22) | 37.0 (7.56) | 36.9 (7.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 100 | 99 | 98 | 394
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 1 | 1 | 5
  Asian | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 19 | 25 | 32 | 23 | 99
  White | 75 | 71 | 65 | 70 | 281
  Other | 0 | 3 | 0 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Weight [Mean (Standard Deviation); unit: Pound] | 164.40 (42.050) | 168.17 (37.867) | 173.97 (43.229) | 179.15 (45.872) | 171.41 (42.532)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 27.73 (6.171) | 28.47 (6.616) | 29.17 (7.096) | 29.92 (7.181) | 28.82 (6.802)
Of Childbearing Potential [Number; unit: Participants]
  Of Childbearing Potential | 72 | 76 | 70 | 65 | 283
  Surgically Sterile | 25 | 24 | 29 | 32 | 110
  Data Missing | 0 | 0 | 0 | 1 | 1
Weight Quartile [Number; unit: Pound]
  95 - 143 pounds | 37 | 21 | 23 | 21 | 102
  >143 - 165 pounds | 18 | 36 | 25 | 24 | 103
  >165 - 200.6 pounds | 23 | 26 | 28 | 24 | 101
  >200.6 - 350 pounds | 19 | 17 | 23 | 28 | 87
  Data Missing | 0 | 0 | 0 | 1 | 1
Menses Frequency [Number; unit: Participants]
  Variable cycle length (<7 days different from nor | 3 | 4 | 4 | 4 | 15
  Regular | 72 | 75 | 86 | 79 | 312
  Variable cycle length (>7 days different from nor | 7 | 2 | 1 | 2 | 12
  2 or more skipped cycles, and amenorrhea for 60 or | 2 | 6 | 2 | 1 | 11
  N.A. | 13 | 13 | 6 | 12 | 44
Natural Hair Color [Number; unit: Participants]
  Red | 6 | 5 | 6 | 6 | 23
  Other Than Red | 91 | 95 | 93 | 92 | 371
Diagnosis [Number; unit: Participants]
  FSAD | 4 | 3 | 3 | 2 | 12
  HSDD | 24 | 20 | 24 | 24 | 92
  Mixed FSAD/HSDD | 69 | 77 | 72 | 72 | 290
Oral Contraceptive Use within 30 Days of Visit 1 [Number; unit: Participants]
  Yes | 12 | 15 | 11 | 15 | 53
  No | 85 | 85 | 88 | 83 | 341

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint is Change From Baseline to End of Study in the Number of Satisfying Sexual Events (SSE)
Description: The primary efficacy endpoint is change from baseline to end of study in the number of satisfying sexual events (SSEs), computed as the number of events during the last 4 weeks of treatment with FSEP-R Q10 = "Yes" minus the number of baseline events with FSEP-R Q10 = "Yes." Efficacy analyses were done with the MITT population which consisted of all randomized subjects who took at least 1 dose of double-blind treatment after the 2 in-clinic doses of double-blind medication and who had at least 1 follow-up visit (Visit 10 or later) to ensure that FSEP-R data were reviewed and confirmed by the investigative site.
Time Frame: 4 - 12 weeks from baseline to end of study (total study duration 20 weeks). Baseline was the 4-week single-blind placebo period.
Measure: Mean (Standard Deviation); unit: SSEs
Arm/Group | Placebo | Bremelanotide Arm 1 | Bremelanotide Arm 2 | Bremelanotide Arm 3
Number analyzed (Participants) | 91 | 87 | 75 | 74
SSEs | 0.2 (2.29) | 0.6 (3.55) | 0.7 (1.81) | 0.8 (2.86)
Statistical Analysis 1: Comparison: Placebo vs Bremelanotide Arm 3; Test type: Superiority or Other; p < 0.05, Van Elteren; Mean Difference (Final Values) = 0.0215, 95% CI 2-sided [0.0 to 1.0], Standard Deviation 2.9
Statistical Analysis 2: Comparison: Placebo vs Bremelanotide Arm 1 vs Bremelanotide Arm 2 vs Bremelanotide Arm 3; Test type: Superiority or Other; p < 0.05, Van Elteren; Mean Difference (Final Values) = 0.0012, 95% CI 2-sided [0.00 to 0.06], Standard Deviation 0.0012

2. Secondary Outcome: Change From Baseline to End-of-Study in Arousal Domain Score From Female Sexual Function Index
Description: The FSFI is brief self-report questionnaire that measures female sexual function. The change from baseline to end of study in the arousal domain were obtained from the FSFI Q3 through Q6. The score range is 0-5. For each of the 2 time points, the score was computed programmatically using the algorithm described by Rosen [6], resulting in a score from 0 (min) to 6 (max).
Time Frame: 4-12 weeks from baseline to end of study (total study duration 20 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Bremelanotide Arm 1 | Bremelanotide Arm 2 | Bremelanotide Arm 3
Number analyzed (Participants) | 91 | 87 | 75 | 74
units on a scale | 0.51 (1.371) | 0.35 (1.457) | 0.71 (1.112) | 1.06 (1.146)
Statistical Analysis 1: Comparison: Placebo vs Bremelanotide Arm 1 vs Bremelanotide Arm 2 vs Bremelanotide Arm 3; Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Final Values) = 0.0496

3. Secondary Outcome: Satisfaction With Arousal as Measured by GAQ Question 1
Description: This is the change in Baseline to End-of-Study in Satisfaction with Arousal as measured by GAQ Question 1. GAQ (Global Assessment Questions) is a questionnaire that evaluates overall satisfaction level experienced while using the study drug. Question 1 is "Compared to the start of the study (prior to taking the study drug), how would you describe your satisfaction with your arousal while using the study drug?" The score range is 1 (very much worse) to 7 (very much better).
Time Frame: 4-12 weeks from baseline to end of study (total study duration 20 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Bremelanotide Arm 1 | Bremelanotide Arm 2 | Bremelanotide Arm 3
Number analyzed (Participants) | 91 | 87 | 75 | 74
units on a scale | 0.4 (1.37) | 0.3 (1.43) | 0.5 (1.46) | 0.9 (1.18)
Statistical Analysis 1: Comparison: Placebo vs Bremelanotide Arm 3; Test type: Superiority or Other; p < 0.05, Van Elteren; Mean Difference (Final Values) = 0.0079, 95% CI 2-sided [0.00 to 1.00]

4. Secondary Outcome: Desire Domain From Female Sexual Function Index
Description: The FSFI is brief self-report questionnaire that measures female sexual function. The change from baseline to end of study in the desire domain were obtained from the FSFI Q1 and Q2. The score range is 1-5. For each of the 2 time points, the score was computed programmatically using the algorithm described by Rosen [6], resulting in a score from 0 (min) to 6 (max).
Time Frame: 4-12 weeks from baseline to end of study (total study duration 20 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Bremelanotide Arm 1 | Bremelanotide Arm 2 | Bremelanotide Arm 3
Number analyzed (Participants) | 91 | 87 | 75 | 74
units on a scale | 0.39 (1.075) | 0.33 (1.093) | 0.55 (0.794) | 0.95 (1.003)
Statistical Analysis 1: Comparison: Placebo vs Bremelanotide Arm 3; Test type: Superiority or Other; p < 0.05, Van Elteren; Mean Difference (Final Values) = 0.0012

5. Secondary Outcome: Satisfaction With Desire as Measured by GAQ Question 2
Description: This is the change in Baseline to End-of-Study in Satisfaction with Desire as Measured by GAQ Question 2. GAQ (Global Assessment Questions) is a questionnaire that evaluates overall satisfaction level experienced while using the study drug. Question 2 is "Compared to the start of the study (prior to taking the study drug), how would you describe your satisfaction with your desire while using the study drug?" The score range is 1 (very much worse) to 7 (very much better).
Time Frame: 4-12 weeks from baseline to end of study (total study duration 20 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Bremelanotide Arm 1 | Bremelanotide Arm 2 | Bremelanotide Arm 3
Number analyzed (Participants) | 91 | 87 | 75 | 74
units on a scale | 0.4 (1.31) | 0.3 (1.32) | 0.8 (1.44) | 0.9 (1.20)
Statistical Analysis 1: Comparison: Placebo vs Bremelanotide Arm 3; Test type: Superiority or Other; p < 0.05, Van Elteren; Mean Difference (Final Values) = 0.0013

6. Secondary Outcome: Quality of Relationship With Partner as Measured by GAQ Question 4
Description: This is the change in Baseline to End-of-Study in Quality of Relationship with Partner as Measured by GAQ Question 4. GAQ (Global Assessment Questions) is a questionnaire that evaluates overall satisfaction level experienced while using the study drug. Question 4 is "Compared to the start of the study (prior to taking the study drug), how has taking the study drug changed your relationship with your partner?" The score range is 1 (very much worse) to 7 (very much better).
Time Frame: 4-12 weeks from baseline to end of study (total study duration 20 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Bremelanotide Arm 1 | Bremelanotide Arm 2 | Bremelanotide Arm 3
Number analyzed (Participants) | 91 | 87 | 75 | 74
units on a scale | 0.3 (1.20) | 0.3 (1.24) | 0.4 (1.22) | 0.6 (1.22)
Statistical Analysis 1: Comparison: Placebo vs Bremelanotide Arm 3; Test type: Superiority or Other; p < 0.05, Van Elteren; Mean Difference (Final Values) = 0.1161

7. Secondary Outcome: FSDS-DAO Total Score
Description: FSDS-DAO (Female Sexual Distress Scale - Desire/Arousal/Orgasm) is an assessment tool to measure female sexual distress. The change from baseline to end of study in the FSDS-DAO (total score) was measured. There are 15 questions, eg, "How often do you feel: Distressed about your sex life" and the score range was 0 (Never), 1 (Rarely), 2 (Occasionally), 3 (Frequently), 4 (Always). The score for each subject at each time point was computed as the sum of the scores from the 15 questions, resulting in a possible score at each time point between 0 and 60.
Time Frame: 4 - 12 weeks from baseline to end of study (total study duration 20 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Bremelanotide Arm 1 | Bremelanotide Arm 2 | Bremelanotide Arm 3
Number analyzed (Participants) | 91 | 87 | 75 | 74
units on a scale | -6.8 (13.57) | -7.4 (13.47) | -9.2 (10.79) | -13.1 (12.93)
Statistical Analysis 1: Comparison: Placebo vs Bremelanotide Arm 3; Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Final Values) = 0.0133

ADVERSE EVENTS:
Arm/Group | Placebo | Bremelanotide Arm 1 | Bremelanotide Arm 2 | Bremelanotide Arm 3
Serious Adverse Events (participants affected / at risk) | 3/97 | 1/100 | 1/99 | 1/98
Other Adverse Events (participants affected / at risk) | 49/97 | 64/100 | 61/99 | 67/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=97) | Bremelanotide Arm 1 (N=100) | Bremelanotide Arm 2 (N=99) | Bremelanotide Arm 3 (N=98)
Escherichia bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=97) | Bremelanotide Arm 1 (N=100) | Bremelanotide Arm 2 (N=99) | Bremelanotide Arm 3 (N=98)
Nausea (Gastrointestinal disorders) | 3 (3) | 18 (34) | 22 (63) | 24 (51)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (6) | 6 (11)
Injection site pain (General disorders) | 3 (6) | 6 (8) | 6 (10) | 7 (9)
Injection site pruritus (General disorders) | 0 (0) | 4 (6) | 4 (7) | 6 (7)
Injection site erythema (General disorders) | 0 (0) | 3 (3) | 3 (5) | 5 (5)
Fatigue (General disorders) | 1 (1) | 3 (4) | 3 (26) | 5 (7)
Injection/vessel puncture site hematoma (1% each) (General disorders) | 1 (1) | 5 (5) | 8 (9) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 9 (10) | 5 (5) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 7 (7) | 8 (8) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 9 (10) | 10 (14) | 15 (18)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 4 (7) | 7 (23)
Paresthesia (Nervous system disorders) | 1 (2) | 2 (3) | 3 (3) | 2 (3)
Flushing (Vascular disorders) | 0 (0) | 17 (36) | 15 (46) | 17 (34)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (4) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 4 (4) | 1 (2)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 3 (5) | 3 (20)
Hypertension (Vascular disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (1) | 3 (3)
Abdominal pain/discomfort, lower/upper abdominal pain, dyspepsia (1% each) (Gastrointestinal disorders) | 2 (2) | 5 (8) | 3 (4) | 4 (7)
Feeling hot/jittery, inj site reac/hemorrhage/rash, pain, chest pain (1% each) (General disorders) | 6 (6) | 5 (8) | 2 (2) | 7 (12)
Fungal infect, gastroenter/bronchitis, vulvo/vaginitis, follicul/pharyngitis, tooth abcess (1% each) (Infections and infestations) | 7 (8) | 7 (8) | 4 (4) | 7 (7)
Migraine, sciatica, sinus headache (1% each) (Nervous system disorders) | 1 (1) | 4 (4) | 3 (3) | 3 (3)
Hematoma, hot flush (1% each) (Vascular disorders) | 1 (1) | 3 (3) | 1 (3) | 3 (3)
Musculoskeletal pain/myalgia, arthralgia, muscle spasms, flank pain (1% each) (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (4) | 3 (3) | 6 (13)
Vag hemorrh/discharge, breast tend/mass, metrorrhagia, menstru irreg, genit discomfort/order (1% ea) (Reproductive system and breast disorders) | 7 (8) | 3 (3) | 4 (4) | 9 (10)
CPK/glu/lipase/chol/BP/triglycerides increased, iron decreased, MCV abnormal (1% each) (Investigations) | 3 (3) | 8 (8) | 4 (4) | 5 (5)
Acne, pruritis, dermatitis contact, erythema, rash, urticaria (1% each) (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (5) | 5 (5) | 3 (3)
Contusion, fall, joint sprain, procedural dizziness/pain, thermal pain (1% each) (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 5 (5) | 4 (4)
Cough, nasal/sinus congestion (1% each) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (7) | 2 (3)
Insomnia, libido increased, restlessness (1% each) (Psychiatric disorders) | 1 (1) | 1 (1) | 4 (22) | 2 (2)
Hypersensitivity, seasonal allergy (1% each) (Immune system disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Melanocytic nevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less